CLINICAL TRIAL: NCT00395655
Title: A Phase II Clinical Study of Hydralazine and Valproic Acid in Combination With Neoadjuvant Cytotoxic Chemotherapy in Stage IIB and IIIA Breast Carcinoma
Brief Title: Hydralazine and Valproate Added to Chemotherapy for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); Psicofarma, S.A. De C.V. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005/012/ICI
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Locally Advanced Breast Cancer
Keywords: locally advanced breast cancer; hydralazine; magnesium valproate; epigenetic therapy; gene expression
MeSH Terms: interventions — Hydralazine

INTERVENTIONS:
Drug: Hydralazine and magnesium valproate administration
Procedure: Core-needle biopsy of the breast

SUMMARY:
Aberrant DNA methylation and histone deacetylation participate in cancer development and progression, as epigenetic alterations are common to breast cancer, in this phase II study, the demethylating hydralazine plus the HDAC inhibitor magnesium valproate will be added to neoadjuvant doxorubicin and cyclophosphamide in locally advanced breast cancer to assess their safety and biological efficacy.

DETAILED DESCRIPTION:
Eligible patients after signing the informed consent and will undergo study evaluation and then typed for acetylator phenotype before being treated with hydralazine at 182 mg for rapid-, or 83 mg for slow-acetylators, and magnesium valproate at 30 mg/kg, starting from day -7 until chemotherapy ends. Chemotherapy will consists in a regimen of four cycles of doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 every 21 days, followed by surgery to assess the pathological response. Adjuvant radiation and additional treatment will be done in off-protocol basis according to standard institutional policies. Blood samples and core-needle biopsies will be taken from primary breast tumors at diagnosis and at day 8 of treatment with hydralazine and valproate. Global cytosine content (global DNA methylation) and histone deacetylase activity will be assessed in peripheral blood DNA. The transcriptional profile in the primary breast tumor before and after treatment will also be analyzed as well as the plasma levels of hydralazine and valproic acid.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 and older; histologically proven invasive T2-3, N0-2, and M0 (stages IIB-IIIA) breast carcinoma; Eastern Cooperative Oncology Group performance status ≤2. Hematological function: Absolute leukocyte count ≥4,000/mm3, platelets ≥100,000/mm3, hemoglobin ≥9.0 g/dL. Hepatic function: total bilirubin, aspartate amino transferase and alanine amino transferase <1.5 the upper normal limit. Renal function: creatinine ≤1.2 mg/dL or a calculated creatinine clearance of ≥60 mL/min. Written informed consent.

Exclusion Criteria:

A history of allergy to sulphas, hydralazine, or magnesium valproate. Past or present condition of rheumatic disease, central nervous system disease, heart failure from aortic stenosis and postural hypotension as diagnosed by a physician. Previous use of the experimental drugs. Pregnancy and breast-feeding. Uncontrolled systemic disease or infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2005-06; Study Completion 2006-08

PRIMARY OUTCOMES:
Global DNA methylation
Histone Deacetylase Activity
Global gene expression

SECONDARY OUTCOMES:
Pathological response
Hydralazine plasma levels
Valproic acid plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Arce, MD, Principal Investigator — Division of Clinical Research, IInstituto Nacional de Cancerologia, Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, TLALPAN, Mexico

REFERENCES:
- [Derived] Arce C, Perez-Plasencia C, Gonzalez-Fierro A, de la Cruz-Hernandez E, Revilla-Vazquez A, Chavez-Blanco A, Trejo-Becerril C, Perez-Cardenas E, Taja-Chayeb L, Bargallo E, Villarreal P, Ramirez T, Vela T, Candelaria M, Camargo MF, Robles E, Duenas-Gonzalez A. A proof-of-principle study of epigenetic therapy added to neoadjuvant doxorubicin cyclophosphamide for locally advanced breast cancer. PLoS One. 2006 Dec 20;1(1):e98. doi: 10.1371/journal.pone.0000098. PMID 17183730